CLINICAL TRIAL: NCT00342355
Title: Randomized, Open-Label 2x2 Factorial Study to Compare the Safety and Efficacy of Different Combination Antiretroviral Therapy Regimens in Treatment Naive Patients With Advanced HIV Disease and/or CD4+ Cell Counts Less Than 200 Cells/MicroL
Brief Title: Antiretroviral Therapy for Advanced HIV Disease in South Africa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Michael Polis, M.D., Michael Polis, National Institute of Allergy and Infectious Diseases (NIAID)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 999904094; 04-I-N094 (Registry Identifier: NCT00342355)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-04

CONDITIONS: HIV
Keywords: Protease Inhibitors; Reverse Transcriptase Inhibitors; AIDS; Opportunistic Infections; Resource-Poor
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opportunistic Infections | interventions — Zidovudine; Stavudine; Didanosine; Lamivudine; efavirenz; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AZT+DDI+EFV (Active Comparator): Zidovudine,Didanosine,Efavirenz ( Zidovudine 600 mg once daily,Didanosine <60 kg/125 mg twice daily or >60kg/200 mg twice daily,Efavirenz 600 mg once daily)
  Interventions: Drug: Zidovudine; Drug: Didanosine; Drug: Efavirenz
- AZT+DDI+r/LPV (Active Comparator): Zidovudine,Didanosine,Lopinavir/Ritonavir(AZT 600 mg once daily,DDI 100 mg twice daily,r/LPV 400mg/100mg twice daily)
  Interventions: Drug: Zidovudine; Drug: Didanosine; Drug: Lopinavir/Ritonavir
- d4T+3TC+EFV (Active Comparator): Stavudine,Lamivudine,Efavirenz(d4T 40 mg twice daily,3TC 300 mg once daily,EFV 600 mg once daily)
  Interventions: Drug: Stavudine; Drug: Lamivudine; Drug: Efavirenz
- d4T+3TC+r/LPV (Active Comparator): Stavudine,Lamivudine,Lopinavir/Ritonavir(d4T 40m mg twice daily,3TC 300 mg once daily,r/LPV 400mg/100mg twice daily)
  Interventions: Drug: Stavudine; Drug: Lamivudine; Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Zidovudine — 600 mg once daily
  Other Names: AZT
  Arms: AZT+DDI+EFV; AZT+DDI+r/LPV
Drug: Stavudine — 40 mg once daily
  Other Names: D4T
  Arms: d4T+3TC+EFV; d4T+3TC+r/LPV
Drug: Didanosine — <60 kg/125 mg twice daily or >60kg/200 mg twice daily
  Other Names: DDI
  Arms: AZT+DDI+EFV; AZT+DDI+r/LPV
Drug: Lamivudine — 300 mg once daily
  Other Names: 3TC
  Arms: d4T+3TC+EFV; d4T+3TC+r/LPV
Drug: Efavirenz — 600 mg once daily
  Other Names: EFV
  Arms: AZT+DDI+EFV; d4T+3TC+EFV
Drug: Lopinavir/Ritonavir — r/LPV 400mg/100mg twice daily
  Other Names: Kaletra
  Arms: AZT+DDI+r/LPV; d4T+3TC+r/LPV

SUMMARY:
This study will determine how well four different antiretroviral drug therapies work in patients with advanced HIV disease. The trial is part of the South Africa-U.S. Project Phidisa Programme - a collaboration between the South African Military Health Service (SAMHS) of the South African National Defense Force (SANDF), the U.S. Department of Defense, and the U.S. National Institutes of Health - to help prevent HIV transmission among South African military and civilian employees and their families.

Members of the SANDF with HIV infection may be eligible for this study. HIV-infected family members who are 14 years of age and older may also participate. All participants must have a CD4 count of less than 200 or an AIDS-defining illness.

Participants are randomly assigned to one of the following four antiretroviral drug regimens, which require taking 5 pills or more every day:

* AZT (zidovudine) + ddl (didanosine) + EFV (efavirenz)
* AZT (zidovudine) + ddl (didanosine) + r/LPV (lopinavir/ritonavir)
* D4T (stavudine) + 3TC (lamivudine) + EFV (efavirenz)
* D4T (stavudine) + 3TC (lamivudine) + r/LPV (lopinavir/ritonavir)

Patients are followed for up to 6 years. Clinic visits are scheduled once a month for the first 3 months and then once every 3 months for the next five years. Patients undergo a medical history, physical examination, and blood tests at each visit, and complete questionnaires of behavior, quality of life, and force readiness every year.

DETAILED DESCRIPTION:
This is a randomized, open label 2x2 factorial study of four regimens of initial therapy.

I. AZT + ddl + EFV

II. AZT + ddl + r/LPV

III. D4T + 3TC + EFV

IV. D4T + 3TC + r/LPV

Eligible patients will commence their randomly allocated study drugs as soon as possible after randomization. Episodes of treatment limiting toxicity will be managed in keeping with protocol specified guidelines.

Patients who experience treatment failures (as specified in the protocol) will be managed by changing their regimen to that corresponding to one of the other treatment groups.

ELIGIBILITY:
* INCLUSION CRITERIA:

Uniformed SANDF personnel or family members of SANDF personnel who are registered as eligible for health services from the SAMHS.

HIV positive as diagnosed and/or confirmed in PHIDISA I OR documented HIV infection from an accredited source.

CD4+ cell count less than 200 cells/microL (or less than or equal to 14% for patients post-splenectomy) AND/OR any AIDS defining illness currently or historically. Patients with pulmonary tuberculosis must have a CD4+ cell count less than 200 cells/microL. Patients with KS must have a CD4+ cell count less than 200 cells/microL unless their sarcoma is progressive and/or requires chemotherapy.

Antiretroviral treatment naive (less than 7 days cumulative exposure to any antiretroviral drug) or treated for post-exposure prophylaxis without becoming HIV infected at that time.

Laboratory variables as follows:

1. Haemoglobin greater than or equal to 9.0g/dL for men and greater than or equal to 8.0g/dL for women.
2. Absolute neutrophil count greater than or equal to 500 cells/microL.
3. Platelet count greater than or equal to 25,000/mm(3).
4. Serum transaminase (ALT or AST) less than or equal to 5 times upper limit of normal (ULN).

   14 years or older.

   Likely to be compliant with study procedures and clinical visits in the opinion of the clinical investigator (guidance is provided in the protocol to assist clinicians in making this decision).

   Have completed the PHIDISA treatment adherence counseling session.

   Provision of written informed consent.

   EXCLUSION CRITERIA:

   Any history of pancreatitis or serious pathology indicative of increased risk for pancreatitis.

   Current requirement for use of a medication that is contra-indicated with the PHIDISA II study drugs. Where possible, alternate therapies should be selected in order to facilitate randomization. Patients entering the study with tuberculosis should defer screening and randomization until successful completion of an induction course of anti-mycobacterium therapy including rifampicin. As appropriate this patient could recommence screening when starting the maintenance regimen of anti-tubercular drugs excluding rifampicin.

   Pregnancy (following delivery, such women may be enrolled).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1771 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Polis, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID); Andrew Ratsela, MD, Principal Investigator — SAMHS
Locations (7):
- South Africa (7):
  - South African Military Health Services (SAMHS), Centurion
  - Umtata Sickbay, Eastaern Cape
  - 3 Military Hospital, Free State
  - 1 Military Hospital, Gauteng
  - Mtubatuba SIckbay, Kwazulu-Natal
  - Phalaborwa Sickbay, Limpopo
  - 2 Military Hospital, Western Cape

REFERENCES:
- [Background] Rabkin M, El-Sadr W, Katzenstein DA, Mukherjee J, Masur H, Mugyenyi P, Munderi P, Darbyshire J. Antiretroviral treatment in resource-poor settings: clinical research priorities. Lancet. 2002 Nov 9;360(9344):1503-5. doi: 10.1016/S0140-6736(02)11478-4. No abstract available. PMID 12433534
- [Background] Hammer SM, Squires KE, Hughes MD, Grimes JM, Demeter LM, Currier JS, Eron JJ Jr, Feinberg JE, Balfour HH Jr, Deyton LR, Chodakewitz JA, Fischl MA. A controlled trial of two nucleoside analogues plus indinavir in persons with human immunodeficiency virus infection and CD4 cell counts of 200 per cubic millimeter or less. AIDS Clinical Trials Group 320 Study Team. N Engl J Med. 1997 Sep 11;337(11):725-33. doi: 10.1056/NEJM199709113371101. PMID 9287227
- [Background] Cameron DW, Heath-Chiozzi M, Danner S, Cohen C, Kravcik S, Maurath C, Sun E, Henry D, Rode R, Potthoff A, Leonard J. Randomised placebo-controlled trial of ritonavir in advanced HIV-1 disease. The Advanced HIV Disease Ritonavir Study Group. Lancet. 1998 Feb 21;351(9102):543-9. doi: 10.1016/s0140-6736(97)04161-5. PMID 9492772
- [Derived] Ledwaba L, Tavel JA, Khabo P, Maja P, Qin J, Sangweni P, Liu X, Follmann D, Metcalf JA, Orsega S, Baseler B, Neaton JD, Lane HC; Project Phidisa Biomarkers Team. Pre-ART levels of inflammation and coagulation markers are strong predictors of death in a South African cohort with advanced HIV disease. PLoS One. 2012;7(3):e24243. doi: 10.1371/journal.pone.0024243. Epub 2012 Mar 20. PMID 22448211
- [Derived] Matthews GV, Manzini P, Hu Z, Khabo P, Maja P, Matchaba G, Sangweni P, Metcalf J, Pool N, Orsega S, Emery S; PHIDISA II study team. Impact of lamivudine on HIV and hepatitis B virus-related outcomes in HIV/hepatitis B virus individuals in a randomized clinical trial of antiretroviral therapy in southern Africa. AIDS. 2011 Sep 10;25(14):1727-35. doi: 10.1097/QAD.0b013e328349bbf3. PMID 21716078
- [Derived] Phidisa II Writing Team for Project Phidisa; Ratsela A, Polis M, Dhlomo S, Emery S, Grandits G, Khabo P, Khanyile T, Komati S, Neaton JD, Naidoo LC, Magongoa D, Qolohle D. A randomized factorial trial comparing 4 treatment regimens in treatment-naive HIV-infected persons with AIDS and/or a CD4 cell count <200 cells/muL in South Africa. J Infect Dis. 2010 Nov 15;202(10):1529-37. doi: 10.1086/656718. Epub 2010 Oct 13. PMID 20942650

RESULTS

PARTICIPANT FLOW:
Groups:
- AZT+ddI+EFV: Zidovudine + Didanosine+Efavirenz
- AZT + ddI + r/LPV: Zidovudine + Didanosine + Lopinavir [LPV] co-formulated with ritonavir [RTV]
- d4T + 3TC + EFV: Stavudine + Lamivudine + Efavirenz
- d4T + 3TC + r/LPV: Stavudine + Lamivudine + lopinavir/ritonavir
Period: Overall Study
Arm/Group | AZT+ddI+EFV | AZT + ddI + r/LPV | d4T + 3TC + EFV | d4T + 3TC + r/LPV
Started | 444 | 440 | 444 | 443
Completed | 444 | 440 | 444 | 443
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZT+ddI+EFV | AZT + ddI + r/LPV | d4T + 3TC + EFV | d4T + 3TC + r/LPV | Total
Number analyzed (Participants) | 444 | 440 | 444 | 443 | 1771
Age Continuous [Mean (Standard Deviation); unit: years] | 35.3 (5.4) | 35.3 (5.4) | 35.5 (5.5) | 35.6 (5.5) | 35.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 135 | 144 | 142 | 567.0
  Male | 298 | 305 | 300 | 301 | 1204.0
Region of Enrollment [Number; unit: participants]
  South Africa | 444 | 440 | 444 | 443 | 1771.0

OUTCOME MEASURES:

1. Secondary Outcome: Serious Adverse Events
Description: Safety outcomes in four different randomly assigned regimens
Time Frame: January 2004 until March 31, 2008
Measure: Number; unit: participant
Arm/Group | AZT+ddI+EFV | AZT + ddI + r/LPV | d4T + 3TC + EFV | d4T + 3TC + r/LPV
Number analyzed (Participants) | 444 | 440 | 444 | 443
participant | 73 | 69 | 64 | 60

2. Primary Outcome: Progression to AIDS or Death in tx naïve Pts With Adv HIV dx in the Four Randomly Assigned Regimens.
Description: Progression of disease, AIDS, or death in treatment naive patients with advanced HIV diagnosis will be evaluated in the four randomly assigned regimens.
Time Frame: January 2004 until March 31 2008
Measure: Number; unit: participants
Arm/Group | AZT+ddI+EFV | AZT + ddI + r/LPV | d4T + 3TC + EFV | d4T + 3TC + r/LPV
Number analyzed (Participants) | 444 | 440 | 444 | 443
participants | 93 | 77 | 70 | 80

ADVERSE EVENTS:
Time Frame: 24.7 months
Arm/Group | AZT+ddI+EFV | AZT + ddI + r/LPV | d4T + 3TC + EFV | d4T + 3TC + r/LPV
Serious Adverse Events (participants affected / at risk) | 96/444 | 85/440 | 72/444 | 71/443
Other Adverse Events (participants affected / at risk) | 0/444 | 0/440 | 0/444 | 0/443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZT+ddI+EFV (N=444) | AZT + ddI + r/LPV (N=440) | d4T + 3TC + EFV (N=444) | d4T + 3TC + r/LPV (N=443)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 12 (12) | 9 (9) | 5 (5) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 21 (21) | 15 (15) | 10 (10) | 15 (15)
General Disorders (General disorders) | 7 (7) | 6 (6) | 7 (7) | 3 (3)
Hepatobilary Disorders (Hepatobiliary disorders) | 3 (3) | 6 (6) | 2 (2) | 3 (3)
Infections and Infestattions (Infections and infestations) | 15 (15) | 15 (15) | 12 (12) | 12 (12)
Injury,poisoning, and procedure complications (Injury, poisoning and procedural complications) | 8 (8) | 4 (4) | 4 (4) | 5 (5)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 15 (15) | 8 (8) | 16 (16) | 15 (15)
Nervous System disorders (Nervous system disorders) | 4 (4) | 5 (5) | 6 (6) | 6 (6)
Psychiatric disorders (Psychiatric disorders) | 7 (7) | 8 (8) | 7 (7) | 3 (3)
Renal and Urinary Disorders (Renal and urinary disorders) | 1 (1) | 4 (4) | 1 (1) | 4 (4)
Vascular disorders (Vascular disorders) | 3 (3) | 5 (5) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No